CLINICAL TRIAL: NCT04950465
Title: An 8 Week, Randomised, Examiner-blind, Controlled Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Dentifrice in the Relief of Dentinal Hypersensitivity in a Chinese Population
Brief Title: A Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Dentifrice in the Relief of Dentinal Hypersensitivity in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 216954
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Apply a full ribbon of toothpaste on the head of the toothbrush provided. Brush teeth for 1*-timed minute, followed by brushing of the qualifying sensitive teeth. Following brushing rinse once with 10 milliliter (ml) of water from the rinsing cup provided.
  Interventions: Other: Sensodyne Sensitivity & Gum
- Negative Control (Active Comparator): Apply a full ribbon of toothpaste on the head of the toothbrush provided; brush teeth for 1* timed minute. Following brushing rinse once with 10 ml of water from the rinsing cup provided.
  Interventions: Other: Crest Cavity Protection Fresh Lime
- Positive Control (Active Comparator): Apply a full ribbon of toothpaste on the head of the toothbrush provided; brush teeth for 1* timed minute. Following brushing rinse once with 10 ml of water from the rinsing cup provided.
  Interventions: Other: Sensodyne Repair and Protect

INTERVENTIONS:
Other: Sensodyne Sensitivity & Gum — Sensodyne Sensitivity & Gum toothpaste containing 0.454% SnF2.
  Arms: Test Dentifrice
Other: Crest Cavity Protection Fresh Lime — Crest Cavity Protection Fresh Lime is containing 1150 parts per million fluoride as Sodium fluoride.
  Arms: Negative Control
Other: Sensodyne Repair and Protect — Sensodyne Repair and Protect dentifrice containing 5.0% weight/weight calcium sodium phosphosilicate.
  Arms: Positive Control

SUMMARY:
The purpose of this study is to support long-term dentinal hypersensitivity (DH) relief claims of 0.454 percent (%) stannous fluoride (SnF2) containing toothpastes in China.

DETAILED DESCRIPTION:
This study will be a single centre, randomised, controlled, examiner-blind, 3 treatment arm, parallel group design study, stratified by maximum baseline Schiff sensitivity score (of the 2 selected 'test teeth'), with a treatment period of 8 weeks, to investigate the clinical efficacy of a SnF2 dentifrice in the reduction of DH in a Chinese population. The SnF2 test dentifrice will be compared to commercialised negative and positive control dentifrices. Participants will be instructed to brush teeth with their assigned dentifrice according to the product use instructions provided. DH assessments will be conducted at Baseline, 4 and 8 weeks. Participants will also be requested to complete a short-form version of the Dentine Hypersensitivity Experience Questionnaire (DHEQ-15) at the Baseline and Week 8 Visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant who presents the following oral and dental inclusions will apply at Screening (Visit 1):

  1. Self-reported history of dentinal hypersensitivity lasting more than six months but not more than 10 years.
  2. Good general oral health, with a minimum of 20 natural teeth.
  3. Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria:

  i. Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR).

ii. Tooth with MGI score ≤1 adjacent to the test area (exposed dentine) only and a clinical mobility of less than or equal to (<=)1.

iii. Tooth with signs of sensitivity measured by a qualifying tactile stimulus (yeaple [<=] 20 gram [g]) and qualifying evaporative air assessment (Schiff sensitivity score more than or equal to (>=) 2).

The following dental inclusions will apply at Baseline (Visit 2):

d) Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), with signs of sensitivity, measured by response to a qualifying tactile stimulus (yeaple <= 20g) and evaporative air assessment (Schiff sensitivity score >=2). The 2 selected 'test teeth' must have also qualified at Screening for this criteria.

- Participant must own a smartphone with the WeChat application installed.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant who has participated in another tooth desensitising treatment study within 8 weeks of the Screening visit.
* A participant with, in the opinion of the investigator or medically qualified designee, has an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant or intending to become pregnant over the duration of the study. This will be confirmed verbally at Screening.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who rinses with water during the first minute of toothbrushing at the Screening visit.
* A participant unwilling or unable to comply with product usage instructions or Lifestyle Considerations that will be described in the protocol.
* A participant with history of regular alcohol and/or substance abuse.
* A participant who has received treatment with another investigational product within 30 days of the first dose of investigational product.
* A participant who has had dental prophylaxis within 4 weeks of Screening, or who requires antibiotic prophylaxis for dental procedures.
* A participant with a tongue or lip piercing.
* A participant with advanced periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* A participant who has had teeth bleaching within 8 weeks of Screening.
* A participant who has used an over-the-counter (OTC) desensitising product (Eg. dentifrice) and/or professional desensitising treatment within 8 weeks of Screening. Participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients.
* A participant with exposed tooth dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel.
* A participant with sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine Eg. current or recent dental caries, or reported treatment of decay within 12 months of Screening.
* A participant who has taken daily doses of medication/treatments or traditional herbal ingredients/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, antidepressants, mood-altering and anti-inflammatory drugs. Examples of herbal ingredients/treatments include clove oil, olive oil, or other treatments that are directly applied to the oral cavity for the treatment of oral health conditions.
* A participant who is taking antibiotics and/or has taken antibiotics within 2 weeks of Screening and/or Baseline.
* A participant who has taken daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — Preventive Dentistry Depart-ment, Shanghai Ninth Peo-ple's Hospital, Shanghai Jiao-tong University, School of Medicine
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Li R, Yang W, Grimaldi R, Zeng P, Smith G, Chen X. Efficacy of a stannous fluoride dentifrice for relieving dentinal hypersensitivity in Chinese population: an 8-week randomized clinical trial. Clin Oral Investig. 2024 Mar 26;28(4):230. doi: 10.1007/s00784-024-05610-9. PMID 38530474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in China.
Pre-assignment Details: A total of 561 participates were screened, out of which 271 participants were enrolled and 197 participates were randomized to a treatment (66 participants in the test product group, 67 participants in the negative control dentifrice group and 64 participants in the positive control dentifrice group) and 196 participants subsequently completed the study; 1 participant did not complete the study from the test product group due to being lost to follow-up.
Groups:
- Test Dentifrice (Sensodyne Sensitivity & Gum): Participants were instructed to brush their teeth for 1 timed minute with full ribbon of toothpaste on the head of the toothbrush provided, followed by brushing of the qualifying sensitive teeth. Following brushing they were instructed to rinse once with 10 milliliters (mL) of water from the rinsing cup provided.
- Negative Control (Crest Cavity Protection Fresh Lime); Positive Control (Sensodyne Repair and Protect): Participants were instructed to brush their teeth for 1 timed minute with full ribbon of toothpaste on the head of the toothbrush provided. Following brushing they were instructed to rinse once with 10 mL of water from the rinsing cup provided.
Period: Overall Study
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime) | Positive Control (Sensodyne Repair and Protect)
Started | 66 | 67 | 64
Completed | 65 | 67 | 64
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population, defined as all participants who are randomized, received at least one dose of the study treatments and provided at least one post-baseline assessment of efficacy.
Groups:
- Test Dentifrice (Sensodyne Sensitivity & Gum): Participants were instructed to brush their teeth for 1 timed minute with full ribbon of toothpaste on the head of the toothbrush provided, followed by brushing of the qualifying sensitive teeth. Following brushing they were instructed to rinse once with 10 mL of water from the rinsing cup provided.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime) | Positive Control (Sensodyne Repair and Protect) | Total
Number analyzed (Participants) | 65 | 67 | 64 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8.04) | 42.7 (8.55) | 42.4 (9.68) | 43.0 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 64 | 56 | 177
  Male | 8 | 3 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 65 | 67 | 64 | 196
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 8 (Test Dentifrice Versus [vs.] Negative Control)
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of 2 selected test teeth, response of participants were scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Higher score indicates worst outcome (more sensitivity). Change from baseline was defined as post dose visit value minus baseline visit value. Baseline was defined as Day 1 (visit 2) value.
Time Frame: Baseline and Week 8
Population: mITT population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 65 | 67
Score on a scale | -0.98 (0.099) | -1.14 (0.098)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity & Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.2639, ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.12 to 0.43], Standard Error of Mean 0.140

2. Secondary Outcome: Change From Baseline in Tactile Threshold at Week 4 and 8 (Test Dentifrice vs. Negative Control)
Description: Constant pressure was administered using Yeaple Probe. At baseline the upper test limit was 20 gram (g) and at Week 4 and 8, the upper test limit was 80g. The tactile threshold was the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth were determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutives 'yes' responses were recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Change from baseline was defined as post dose visit value minus baseline visit value. Baseline was defined as Day 1 (visit 2) value.
Time Frame: Baseline, Week 4 and 8
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 65 | 67
grams
  Week 4: number analyzed (Participants) | 64 | 67
  Week 4 | 9.22 (1.577) | 7.42 (1.538)
  Week 8 | 16.63 (2.393) | 11.82 (2.353)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity & Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 4; Test type: Superiority; p = 0.6978, Van Elteren Test; Due to non-normal residual analyses from ANCOVA a Van Elteren Test was performed
Statistical Analysis 2: Comparison: Test Dentifrice (Sensodyne Sensitivity & Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 8; Test type: Superiority; p = 0.8130, Van Elteren Test; Due to non-normal residual analyses from ANCOVA a Van Elteren Test was performed

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 4 (Test Dentifrice vs. Negative Control)
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of 2 selected test teeth, response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Higher score indicates worst outcome (more sensitivity). Change from baseline was defined as post dose visit value minus baseline visit value. Baseline was defined as Day 1 (visit 2) value.
Time Frame: Baseline and Week 4
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 64 | 67
Score on a scale | -0.79 (0.082) | -0.75 (0.080)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity & Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.7645, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.26 to 0.19], Standard Error of Mean 0.115

4. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 4 and 8 (Positive Control vs. Negative Control)
Description: as for outcome 3
Time Frame: Baseline, Week 4 and Week 8
Population: mITT population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 64 | 67
score on a scale
  Week 4 | -0.76 (0.082) | -0.75 (0.080)
  Week 8 | -0.99 (0.100) | -1.14 (0.098)
Statistical Analysis 1: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 4; Test type: Superiority; p = 0.9728, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.23 to 0.22], Standard Error of Mean 0.114
Statistical Analysis 2: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 8; Test type: Superiority; p = 0.2968, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.13 to 0.42], Standard Error of Mean 0.140

5. Secondary Outcome: Change From Baseline in Tactile Threshold at Week 4 and 8 (Positive Control vs. Negative Control)
Description: Constant pressure was administered using Yeaple Probe. At baseline the upper test limit was 20g and at Week 4 and 8, the upper test limit was 80g. The tactile threshold was the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutives 'yes' responses would be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Change from baseline was defined as post dose visit value minus baseline visit value. Baseline was defined as Day 1 (visit 2) value.
Time Frame: Baseline, Week 4 and Week 8
Population: mITT population
Measure: Mean (Standard Error); unit: grams
Arm/Group | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 64 | 67
grams
  Week 4 | 4.59 (1.577) | 7.42 (1.538)
  Week 8 | 11.05 (2.412) | 11.82 (2.353)
Statistical Analysis 1: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 4; Test type: Superiority; p = 0.1682, Van Elteren Test; Due to non-normal residual analyses from ANCOVA a Van Elteren Test was performed
Statistical Analysis 2: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Week 8; Test type: Superiority; p = 0.3937, Van Elteren Test; Due to non-normal residual analyses from ANCOVA a Van Elteren Test was performed

ADVERSE EVENTS:
Time Frame: From start of screening until end of study (up to Day 57+/-3)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) is a particular category of an adverse event where the adverse outcome is serious.
Arm/Group | Test Dentifrice (Sensodyne Sensitivity & Gum) | Negative Control (Crest Cavity Protection Fresh Lime) | Positive Control (Sensodyne Repair and Protect)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 18/66 | 3/67 | 10/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (Sensodyne Sensitivity & Gum) (N=66) | Negative Control (Crest Cavity Protection Fresh Lime) (N=67) | Positive Control (Sensodyne Repair and Protect) (N=64)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (Sensodyne Sensitivity & Gum) (N=66) | Negative Control (Crest Cavity Protection Fresh Lime) (N=67) | Positive Control (Sensodyne Repair and Protect) (N=64)
Dental abfraction (Gastrointestinal disorders) | 4 | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Angular cheilitis (Gastrointestinal disorders) | 2 | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 3 | 0 | 0
Oral blood blister (Gastrointestinal disorders) | 1 | 0 | 1
Gingival erythema (Gastrointestinal disorders) | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04950465/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04950465/SAP_001.pdf